CLINICAL TRIAL: NCT00598936
Title: A Prospective Study With a New Device for the Monitoring of Cerebral Oxygenation on Cardiac Surgery Patients
Status: Terminated | Type: Observational
Why Stopped: Investigator considered the device with no clinical utility.
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-5840
Record Dates: First submitted 2007-12-24; First posted 2008-01-23 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Artery Disease; Heart Valve Disease
Keywords: Hypoxia; Cerebral Hypoxia
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Hypoxia; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac Surgery or Hospitalization: Patients scheduled for a Cardiac Surgery procedure, two types of cerebral oximetry devices were compared at the same time during the surgical procedure.
  The second group were patients hospitalized (in the Intensive Care Unit or ICU, with any diagnosis, excluding head trauma patients. Those patients were monitored using two types of cerebral oximetry devices at the same time for up to 72 hours.
  Interventions: Device: CDI 1000 COM and INVOS 5100

INTERVENTIONS:
Device: CDI 1000 COM and INVOS 5100 — CDI 1000 and INVOS 5100 sensors were attached to subject's forehead for a 12 hour period, digital photographs were taken before and after sensor placement.
  Other Names: Terumo CDI 1000 COM; Somanetics INVOS 5100

SUMMARY:
The purpose of this study is to determine whether a new cerebral oxygenation monitoring device is comparatively similar to the current approved devices.

DETAILED DESCRIPTION:
Cerebral oxygenation monitoring is an innovative way to monitoring cardiac surgery patients intraoperatively to reduce the incidence of postoperative hypoxic side effects. There are a number of approved devices already in the market that have proved their efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. To be 18 years old or older
2. Scheduled for cardiac surgery
3. Treatment will include 72 hours or more of hospital stay
4. Understand enough about the risks and benefits of the study to be able to make an informed decision before agreeing to be in the study

Exclusion Criteria:

1. History of cerebrovascular disease
2. History of skin problems on forehead (skin rashes, acne, allergies, etc.)
3. History of craniofacial surgeries
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects ≥18 year-old of age admitted to the University Hospital setting scheduled for cardiac surgery or admitted for any cause to the Intensive Care Unit (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To test a new device for Cerebral Oxygenation Monitoring | 12 hours

SECONDARY OUTCOMES:
Safety of human forehead skin during period of probe adhesion | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Milliken, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States